CLINICAL TRIAL: NCT04002128
Title: Tracheal Colonization and Outcome After Major Abdominal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osijek University Hospital (Other)
Collaborators: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 01
Record Dates: First submitted 2019-06-24; First posted 2019-06-28 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Neoplasms Malignant; Surgical Procedures, Operative; Stomach Neoplasms; Pancreatic Cancer, Adult
Keywords: tracheal colonization;; Bacteria;; Survival; Anesthesia, General;
MeSH Terms: conditions — Colonic Neoplasms; Stomach Neoplasms; Pancreatic cancer, adult

STUDY DESIGN:
Intervention Model Description: To investigate whether productive cough, dyspnea and hoarseness were different between two groups of patients. Group Air received sevoflurane anesthesia with 35% O2 in air, and Group N2O received sevoflurane anesthesia with 35% O2 in N2O
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Postoperative outcomes were registered by doctor who did not know type of anesthesia delivered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group air (Placebo Comparator): Group air was mechanically ventilated using 35% oxygen in 65% air during the whole surgical procedure.
  Thiopental sodium was used for induction of anesthesia, muscle relaxation was maintained with vecuronium. General anesthesia with sevoflurane was maintained during the surgical procedure. Intraoperative analgesia was achieved with fentanyl boluses.
  Interventions: Other: Tracheal aspirates and nasal smears were taken in all the patients. Laparotomies were performed in all patients.
- Group nitrous oxyde (N2O) (Active Comparator): Group N2O was mechanically ventilated using 35 % oxygen and 65 % of nitrous oxyde during the surgical procedure.
  Nitrous oxyde may increase cuff pressure during the general endotracheal anesthesia and result in the respiratory symptoms like sore throat, hoarseness and postoperative cough.
  Thiopental sodium was used for induction of anesthesia, muscle relaxation was maintained with vecuronium. General anesthesia with sevoflurane was maintained during the surgical procedure. Intraoperative analgesia was achieved with fentanyl boluses.
  Interventions: Other: Tracheal aspirates and nasal smears were taken in all the patients. Laparotomies were performed in all patients.

INTERVENTIONS:
Other: Tracheal aspirates and nasal smears were taken in all the patients. Laparotomies were performed in all patients. — Nitrous oxyde and sevoflurane anesthesia may alter mucus transport in the early postoperative period. In colonized patients it may result in more respiratory complications.

SUMMARY:
The goals of this study were to investigate whether two anesthesia regimens, with and without N2O, and bacterial colonization influence respiratory complications after major abdominal surgery for cancer.

DETAILED DESCRIPTION:
A study was approved by institutional ethics committee. All patients were informed on the study protocol by attending anesthesiologist on the day of the surgery and written informed consent was obtained. Patients with clinically or radiologically confirmed acute respiratory infections or those using antibiotics due to the respiratory infections a week prior to the surgery were not included in the study. Following risk factors were recorded in all patients: age, sex, weight loss in the last 6 months, comorbidities and operative time. Comorbidities were rated using ASA status and Charlson comorbidity index by 3 independent observers. Charlson comorbidity index was calculated after pathological examination. An advanced malignant disease was considered if tumor had infiltrated other organs or surrounding tissues, or when positive lymph nodes or metastases were confirmed.

A group of 120 colorectal, gastric, or pancreatic cancer patients scheduled for surgery in the single centre were included in the prospective randomized study regardless of their ASA physical status. Nasopharyngeal smears were obtained in the preoperative area and tracheal aspirates were obtained in the operating room at the end of the surgery with a sterile suction catheter in a closed system.

Postoperative Hgb; CRP and lung auscultation were done in all patients on the second and fourth postoperative day.

Outcome measures registered were:

* Postoperative pneumonia
* Productive and difficult cough
* Dysphonia
* Congestive heart failure
* postoperative complications, including hypertensive crisis, thromboembolic and infective complications were summarized one year after surgical treatment was finished & one year survival

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosis of gastric cancer, or colorectal cancer or pancreatic cancer
* Scheduled for major abdominal surgery with organ resections
* Written informed consent
* Nasopharyngeal smears taken in the preoperative area
* Tracheal aspirates taken at the end of the surgical procedure

Exclusion Criteria:

* Patients unable to understand study protocol and patients who refused study participation at any time
* patients with clinically or radiologically confirmed acute respiratory infections at admission
* antibiotic therapy due to the respiratory infections a week prior to the surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of the patients with postoperative pneumonia | Postoperative day 4
  Number of patients who reported the presence of cough, dyspnea and/or abnormal findings on lung examination, and two of following: fever, leukocytosis or high CRP, and positive chest radiograms.
Number of the patients with productive cough and difficult expectoration | Postoperative day 4
  patients without auscultatory findings who self reported that they have productive sputum and painful expectoration without laboratory and RTG findings suggestive for pneumonia
Number of the patients with hoarseness | Postoperative day 4
  The patients who self-reported hoarseness and changed voice

SECONDARY OUTCOMES:
One year survival and complications | One postoperative year
  All the other postoperative complications, including in-hospital hypertensive crisis, thromboembolic and infective complications were summarized one year after surgical treatment was finished.

CONTACTS AND LOCATIONS:
Overall Officials: Slavica Kvolik, MD, PhD, Principal Investigator — Osijek University Hospital, J. Huttlera 4, 31 000 Osijek, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Upon the request all blinded individual participant data (IPD) may be available to other researchers
Supporting Information: CSR
Time Frame: Upon the request
Access Criteria: Shared by principal investigator directly

REFERENCES:
- [Background] Evaristo-Mendez G, Rocha-Calderon CH. [Risk factors for nosocomial pneumonia in patients with abdominal surgery]. Cir Cir. 2016 Jan-Feb;84(1):21-7. doi: 10.1016/j.circir.2015.05.051. Epub 2015 Aug 8. Spanish. PMID 26259742
- [Background] Fernandez-Bustamante A, Frendl G, Sprung J, Kor DJ, Subramaniam B, Martinez Ruiz R, Lee JW, Henderson WG, Moss A, Mehdiratta N, Colwell MM, Bartels K, Kolodzie K, Giquel J, Vidal Melo MF. Postoperative Pulmonary Complications, Early Mortality, and Hospital Stay Following Noncardiothoracic Surgery: A Multicenter Study by the Perioperative Research Network Investigators. JAMA Surg. 2017 Feb 1;152(2):157-166. doi: 10.1001/jamasurg.2016.4065. PMID 27829093
- [Background] de Albuquerque Medeiros R, Faresin S, Jardim J. [Postoperative lung complications and mortality in patients with mild-to-moderate COPD undergoing elective general surgery]. Arch Bronconeumol. 2001 May;37(5):227-34. doi: 10.1016/s0300-2896(01)75059-4. Spanish. PMID 11412514
- [Background] Payne KA, Miller DM. The Miller tracheal cuff pressure control valve. Clinical use in controlled and spontaneous ventilation. Anaesthesia. 1993 Apr;48(4):324-7. doi: 10.1111/j.1365-2044.1993.tb06954.x. PMID 8494136
- [Background] Braz JR, Volney A, Navarro LH, Braz LG, Nakamura G. Does sealing endotracheal tube cuff pressure diminish the frequency of postoperative laryngotracheal complaints after nitrous oxide anesthesia? J Clin Anesth. 2004 Aug;16(5):320-5. doi: 10.1016/j.jclinane.2004.03.001. PMID 15374551